CLINICAL TRIAL: NCT01262937
Title: A Pilot Study to Examine the Human Gastrointestinal Tract Using the Confocal Endomicroscope
Brief Title: A Study to Examine the Human Gastrointestinal Tract Using the Confocal Endomicroscope
Status: Terminated | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0706002810
Record Dates: First submitted 2010-12-14; First posted 2010-12-20 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Digestive System Diseases
Keywords: confocal, biliary, esophagus
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Biliary Confocal Imaging
  Interventions: Device: Confocal Imaging
- Esophageal Confocal Imaging
  Interventions: Device: Confocal Imaging

INTERVENTIONS:
Device: Confocal Imaging — Confocal imaging performed of the digestive system with the use of confocal miniprobes such as the Gastroflex UHD and Cholangioflex miniprobes (Cellvizio, Mauna Kea, Paris, France)

SUMMARY:
The goal of the project is to determine whether confocal endomicroscopy can be used to identify and discriminate among dysplastic, neoplastic, and nonneoplastic tissue, as compared with histologic specimens as a reference. The project will evaluate those at risk for or with known Barrett's esophagus, and those with known or suspected biliary strictures. It is our hypothesis that we will be able to identify between neoplastic and nonneoplastic tissue.

DETAILED DESCRIPTION:
This study was amended from it's initial design to increase the number of patients to 200. The study was terminated in July 2016 after 106 patients were enrolled and had completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with long-standing reflux symptoms, undergoing surveillance for Barrett's esophagus, or scheduled for endoscopic therapy with esophageal dysplasia
* Patients undergoing ERCP for known or suspected biliary strictures.

Exclusion Criteria:

* have a known allergy or have had a prior adverse reaction to fluorescent contrast agents or chromoendoscopy stains
* are younger than age 18 or who are mentally or legally incapacitated or unable to give informed consent
* are pregnant or breastfeeding
* patients with advanced esophageal cancer
* acute gastrointestinal bleeding
* coagulopathy
* impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long-standing reflux symptoms, undergoing surveillance for Barrett's esophagus, or scheduled for endoscopic therapy with esophageal dysplasia. Also, patients undergoing ERCP for known or suspected biliary strictures.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To compare confocal image characteristics between benign and malignant tissue. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nathanson, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States